CLINICAL TRIAL: NCT00004350
Title: Evaluation of Fanconi Syndrome and Cystinosis
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of California, San Diego (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Other Study IDs: 199/11911; UCSD-012
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-12

CONDITIONS: Cystinosis; Fanconi Syndrome
Keywords: Fanconi syndrome; cystinosis; rare disease; renal and genitourinary disorders
MeSH Terms: conditions — Cystinosis; Fanconi Syndrome; Rare Diseases; Urogenital Diseases

SUMMARY:
OBJECTIVES:

I. Classify renal tubular defects using clinical and biochemical findings in patients with Fanconi syndrome and cystinosis.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Patients receive a clinical and biochemical evaluation, including a psychometric assessment and molecular, renal, and thyroid studies.

ELIGIBILITY:
* Inherited renal tubular defects, i.e., Fanconi syndrome
* Fanconi syndrome due to cystinosis eligible

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12
Dates: Start 1999-10

CONTACTS AND LOCATIONS:
Overall Officials: Jerry A. Schneider, Study Chair — University of California, San Diego